CLINICAL TRIAL: NCT00754286
Title: A Randomized Trial of The Effectiveness of Aromatherapy on Chemotherapy Induced Nausea and Vomiting in Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Soothing Scents, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 08-01-017
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Brain Tumors; Leukemia; Sarcomas; Neuroblastoma; Lymphoma; Hodgkins Disease
Keywords: Aromatherapy
MeSH Terms: conditions — Brain Neoplasms; Leukemia; Sarcoma; Neuroblastoma; Lymphoma; Hodgkin Disease | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aromatherapy (Experimental): Participants will be given aromatherapy wand at the onset of their chemotherapy treatment.
  Interventions: Other: Aromatherapy Scented Wand
- Placebo (Placebo Comparator): Participants will be given the placebo wand at the onset of their chemotherapy treatment. Placebo wands will look identical to the scented wands but will not contain a scent.
  Interventions: Other: Placebo wand

INTERVENTIONS:
Other: Aromatherapy Scented Wand — The aromatherapy used in this will be Quease Ease™, manufactured by Soothing Scents, Inc. Quease Ease is a blend of lavender, spearmint, ginger, and peppermint soaked into a pad placed within a "wand" dispenser that emits a fragrance when placed within a few inches of the nares. Participants will be given aromatherapy wand at the onset of their chemotherapy treatment. Participants will be instructed how to self-administer the aromatherapy treatment. Specifically, they can hold the wand under their nose and breathe in deeply five times when they feel symptoms of nausea or anxiety.
  Other Names: Soothing Scents, Inc.; Quease Ease™; Aromatherapy
  Arms: Aromatherapy
Other: Placebo wand — Placebo wands will look identical to the scented wands but will not contain a scent. Participants will be given the placebo wand at the onset of their chemotherapy treatment. Participants will be instructed how to self-administer the placebo treatment. Specifically, they can hold the wand under their nose and breathe in deeply five times when they feel symptoms of nausea or anxiety.
  Arms: Placebo

SUMMARY:
Aromatherapy has anecdotally been reported to decrease nausea and vomiting, decrease anxiety and increase quality of life in cancer patients. Therefore, the proposed study aims to assess the effectiveness of aromatherapy versus placebo on nausea, vomiting, anxiety and quality of life among pediatric oncology patients receiving emetogenic chemotherapy.

DETAILED DESCRIPTION:
Nausea and vomiting remain two of the most distressing symptoms to children being treated for cancer. Nausea and vomiting are directly associated with the administration of chemotherapy, due to effects of the chemotherapy on the gastrointestinal mucosa, and certain chemotherapeutic agents, such as cisplatin, are known to be particularly emetogenic. In addition, anticipatory anxiety has been identified as an important patient factor in the development of post-chemotherapy nausea and vomiting. Many drugs have been developed in an effort to diminish nausea and vomiting in children receiving emetogenic chemotherapy and these agents, particularly the 5-hydroxytryptamine receptors, have vastly reduced the amount of nausea and vomiting experienced in this population. However, approximately 50% of children and adolescents still suffer from nausea and/or vomiting even after maximal pharmacological intervention. This suggests that other interventions are needed to further reduce the experienced nausea and vomiting seen in children undergoing chemotherapy. As such, many patients and providers have turned to complementary and alternative medicine (CAM) for the relief of nausea and vomiting. Aromatherapy is one such modality that has demonstrated some degree of effectiveness in adults suffering from nausea and vomiting due to chemotherapy, motion sickness, or postoperatively.

Aromatherapy is an inexpensive and easy therapy to administer to children, and many children can self administer aromatherapy depending on their age and the form of aromatherapy. Aromatherapy has anecdotally been reported to decrease nausea and vomiting, decrease anxiety and increase quality of life in cancer patients. Therefore, the proposed study aims to assess the effectiveness of aromatherapy versus placebo on nausea, vomiting, anxiety and quality of life among pediatric oncology patients receiving emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 7-21 with a diagnosis of cancer and will be receiving emetogenic chemotherapy.

Exclusion Criteria:

* Patients allergic to peppermint, ginger or lavender

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Examine the effect of aromatherapy on nausea and vomiting among pediatric oncology patients undergoing chemotherapy. | One week after completed chemotherapy

SECONDARY OUTCOMES:
Effects on anxiety, depression and quality of life in this population | At beginning and at end of chemotherapy cycle

CONTACTS AND LOCATIONS:
Overall Officials: Karen Moody, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States